CLINICAL TRIAL: NCT06195683
Title: Prospective, Single-center, Single-arm Phase 2 Clinical Study on the Efficacy and Safety of Single-agent Neoadjuvant Therapy With Serplulimab in Patients With Non-small Cell Lung Cancer With TPS ≥ 50%.
Brief Title: Serplulimab for Patients With Non-small Cell Lung Cancer (NSCLC) With TPS ≥ 50%: a Prospective, Single-center, Single-arm Phase 2 Study.
Acronym: NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, liujinshi, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-1067 (IIT); IRB-2023-1067 (IIT) (Other: Zhengjiang cancer hospital)
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer; PDL1 Gene Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Participants with ⅠB(≥4cm)-ⅢA and TPS ≥ 50% non-small cell lung cancer patients, excluding EGFR and ALK gene mutations. They will receive 4 cycles of Serplulimab monotherapy at 4.5mg/kg as neoadjuvant treatment before surgery. Subsequently, they will undergo surgical resection and the effectiveness of the neoadjuvant treatment will be evaluated. After surgery, they will receive 14 cycles of Serplulimab as adjuvant treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-PDL-1 Immunotherapy followed by Surgical Resection (Experimental): Participants will receive four preoperative doses of PDL-1 inhibitor Serplulimab in adults with untreated, surgically resectable early (stage IB, II, or IIIA) NSCLC. Serplulimab (at a dose of 4.5mg per kilogram of body weight) was administered intravenously every 3 weeks, with surgery planned approximately 4 weeks after the last dose.
  Interventions: Drug: Serplulimab

INTERVENTIONS:
Drug: Serplulimab — Serplulimab for 4.5mg/kg IV Q3W day 1,22,43,64

SUMMARY:
The goal of this clinical trial is to observe the efficacy and safety of Serplulimab monotherapy as a neoadjuvant treatment for TPS ≥ 50% non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
The study aims to explore new strategies for neoadjuvant treatment of resectable NSCLC patients with TPS ≥ 50%, and to identify potential prognostic biomarkers.

Participants with stage ⅠB-ⅢA and TPS ≥ 50% non-small cell lung cancer, excluding EGFR and ALK gene mutations will receive 4 cycles of Serplulimab monotherapy at 4.5mg/kg as neoadjuvant treatment before surgery. Subsequently, they will undergo surgical resection and evaluation of the effect of neoadjuvant therapy. 14 cycles of Serplulimab as adjuvant treatment. Participants will provide blood samples before neoadjuvant treatment, before the third cycle of neoadjuvant treatment, before surgery, and 4-7 days after surgery for Minimal Residual Disease（MRD） detection to assist in evaluating the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

Sign written informed consent

* The participant signs and dates a written informed consent form. The informed consent form must be signed before any protocol-related procedures (not part of the participant's routine medical care) are performed.
* The participant must be willing and able to comply with scheduled visits, treatment regimens, and laboratory tests.

Participant types and target disease characteristics

-Eastern Cooperative Oncology Group (ECOG) performance status score 0-1 Histologically confirmed non-small cell lung cancer, clinical stage IIB (tumors ≥4cm), II, IIIA (lymph nodes limited to N1) according to the UICC lung cancer staging system (8th edition).

There are measurable lesions according to RECIST criteria.

* Participants must have tumor tissue samples available for PD-L1 (22c3 kit) IHC testing, with PD-L1 expression ≥50%
* Within 3 months, lung function should reach at least FEV1>1.0L, FEV1%>40%.

According to the definition of laboratory test results described below, there is sufficient hematology and vital organ function, and the test results need to be completed within 14 days before the first study treatment:

1. Blood routine (within 14 days before the first study treatment without receiving hematopoietic stimulating factors or blood transfusions): absolute neutrophil count (ANC) ≥ 1.5 × 109/L, absolute lymphocyte count (LC) ≥ 0.5 × 109/L; platelet count (PLT) ≥ 100 × 109/L, hemoglobin (Hb) ≥ 90g/L
2. Liver function: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 xULN; total bilirubin (TBIL) ≤1.5 x ULN (for patients with confirmed Gilbert syndrome, total bilirubin ≤3.0 mg/dL); albumin (ALB) ≥3 g/dL;
3. Renal function: creatinine clearance rate (CrCl) ≥45mL/minute (using the Cockcroft-Gault formula);
4. Coagulation function: international normalized ratio (INR) ≤1.5, activated partial thromboplastin time (APTT) ≤1.5 x ULN;
5. Cardiac color Doppler ultrasound examination: left ventricular ejection fraction (LVEF) ≥50% Age and fertility status Age ≥18 and ≤75. Women of childbearing age (WOCBP) must have a negative serum or urine pregnancy test within 24 hours before starting the study treatment (the minimum sensitivity of HCG is 25 IU/L or equivalent units).

   * Female must be in a non-lactating state

Exclusion Criteria:

Histologically or cytologically confirmed mixed SCLC and NSCLC, large cell neuroendocrine carcinoma, and sarcomatoid carcinoma; NSCLC non-squamous histological type with EGFR mutation-positive or ALK-positive subjects. Non-squamous subjects must undergo EGFR gene testing and ALK gene and/or immunohistochemical testing, with TPS score <50%; Malignant pleural effusion. If the subject has pleural effusion that can be aspirated during the screening period, at least one pleural puncture is required to confirm the presence of malignant cells; Previous systemic treatment for non-small cell lung cancer (including clinical study medication) has been received. If the subject has previously received traditional Chinese medicine for anti-tumor treatment, the end of the treatment must be separated from the first study medication by a time interval of no less than 2 weeks; Previous thoracic radiotherapy has been received; Participation in other clinical studies within 4 weeks before the first dose or 5 half-lives of the study drug, whichever is shorter; Systemic immune stimulation therapy (including but not limited to interferon or interleukin-2, including immune stimulation agents in clinical trials) within 4 weeks before the first dose; Systemic immunosuppressive therapy (including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, thalidomide, antineoplastic cytokines) within 2 weeks before the first dose or is expected to be required during the study treatment period. Subjects who have received short-term, low-dose (≤10mg/day prednisone or equivalent dose) systemic immunosuppressive drugs or short-term high-dose systemic immunosuppressive drugs (such as for treatment of contrast agent allergy with glucocorticoids for 48 hours) may be included in the study after obtaining approval from the medical monitor. Subjects who use glucocorticoids (≤10mg/day prednisone or equivalent dose) for treatment of chronic obstructive pulmonary disease, mineralocorticoids for treatment of orthostatic hypotension, and physiological replacement doses of glucocorticoids for treatment of adrenal insufficiency may be included; There are autoimmune diseases. The following conditions are allowed: type I diabetes (blood sugar can be controlled by insulin therapy); hypothyroidism caused by autoimmune thyroiditis that only needs hormone replacement therapy; only vitiligo dermatosis (psoriatic arthritis needs to be excluded); History of other malignancies (except non-small cell lung cancer) within the screening period, excluding cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostatic cancer, ductal carcinoma in situ, hormone replacement therapy for non-metastatic prostate cancer or breast cancer; Known or suspected interstitial pneumonia or other serious lung diseases that may interfere with lung toxicity testing or treatment, including significant respiratory function impairment; Severe cardiovascular diseases such as NYHA classification II or higher, myocardial infarction or cerebrovascular accident (stroke, hemorrhagic stroke) within 3 months before the first dose, unstable arrhythmia or unstable angina within 1 month before the first dose; Significant bleeding symptoms or bleeding tendency within 1 month before the first dose, such as gastrointestinal bleeding, gastric ulcer bleeding, or suffering from thromboangiitis obliterans; Deep venous thrombosis and pulmonary embolism within 3 months before the first dose; HIV positive; Active hepatitis B (HBsAg positive and HBV-DNA test result higher than the upper limit of normal in the local laboratory during screening) or hepatitis C (HCV-Ab positive and HCV-RNA positive during screening); Active tuberculosis infection within 1 year before the first dose; Serious infection within 4 weeks before the first dose, including hospitalization and/or antibiotics treatment for ≥2 weeks for infections such as sepsis, severe pneumonia, etc.; antibiotics treatment for active infections within 2 weeks before the study treatment; Vaccination with live attenuated vaccines within 28 days before the first dose; Major surgery within 28 days before the first dose; Previous or planned allogeneic bone marrow transplantation or solid organ transplantation; History of severe allergic reaction to other monoclonal antibody / fusion protein drugs; Allergic to any component of the investigational product; Pregnant, breastfeeding, or planning to become pregnant during the study period; Subjects with a history of substance abuse, alcoholism, or drug addiction; The researchers believe that any other medical (such as pulmonary, metabolic, endocrine, or neurological diseases, congenital diseases, etc.), psychiatric, or social conditions that may interfere with the rights, safety, health, or ability of the subjects to sign informed consent, collaborate and participate in the study, or interfere with the evaluation of study drugs, interpretation of patient safety, or study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate, pCR | Assessed 1 month after surgery
Major Pahological Response, MPR | Assessed 1 month after surgery
Objective Response Rate (ORR) | From the time of enrollment, assessed up to 5 years follow-up.
  Proportion of patients with complete response (CR) or partial response (PR) to preoperative multimodal therapy. ORR will be evaluated using RESIST1.1 by CT of the chest.

SECONDARY OUTCOMES:
Overall survival (OS) | From the time of enrollment, assessed up to 5 years follow-up.
  The time from enrollment to death due to any reason. The time from enrollment to death due to any reason. The time from enrollment to death due to any reason.
Event-Free Survival(EFS) | From the time of enrollment, assessed up to 5 years follow-up.
  The time from enrollment to disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No